CLINICAL TRIAL: NCT06425835
Title: Virtual Reality in the Management of Painful or Anxiety-provoking Procedures in Emergency Departments: (Open Prospective Observational Study)
Brief Title: Virtual Reality in the Management of Painful or Anxiety-provoking Procedures in Emergency Departments
Acronym: VR
Status: Not yet recruiting | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, PROFESSOR, University of Monastir
Other Study IDs: UMonastir2024
Record Dates: First submitted 2024-03-14; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Pain and Anxiety; Dislocation; Suture
MeSH Terms: conditions — Pain; Anxiety Disorders; Joint Dislocations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: VR device — The VR device consists of a pair of VR glasses with a video previously chosen and installed. Patient preparation must be done before initiating the protocol.
  The first step is to choose patient candidates for VR who are understanding and interested. Guardian approval is required; then it is necessary to explain the principle, the stages and the benefits of the care.
  The intensity of pain is calculated according to the visual analog scale before, during the procedure and 30 minutes after as well as the max VAS during the procedure, the 'Children Fear Scale', the satisfaction score and any adverse effects are noted.

SUMMARY:
Study and evaluate the effectiveness of virtual reality in pain management.

DETAILED DESCRIPTION:
Study and evaluate the effectiveness of virtual reality in pain management.This is an open prospective observational study carried out at Urgences Fattouma Bourgiba Monastir.

For all patients included, a data collection form must be completed, mentioning age, sex, medical and surgical history, and the type of procedure planned.

* If initial VAS >5 and intolerable: patients will immediately use painkillers and will be excluded from the study.
* If initial VAS <=5 or > 5 but tolerable: Only VR glasses are used as an analgesic.

If during the procedure the patient describes intolerable pain: the VAS will be noted, and the patient will use a rescue analgesic (intranasal ketamine or other at the discretion of the attending physician).

The VR device consists of a pair of VR glasses with a video previously chosen and installed. Patient preparation must be done before initiating the protocol.

The first step is to choose patient candidates for VR who are understanding and interested. Guardian approval is required; then it is necessary to explain the principle, the stages and the benefits of the care.

The intensity of pain is calculated according to the visual analog scale before, during the procedure and 30 minutes after as well as the max VAS during the procedure, the 'Children Fear Scale', the satisfaction score and any adverse effects are noted.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 09 and 24 years
* suturing a wound
* changing a dressing
* lumbar puncture,
* peripheral venous line
* blood test
* intramuscular injection
* reduction of a fracture
* casting or plastering.

Exclusion Criteria:

* impaired consciousness
* epilepsy
* wound/infection covering the helmet area
* headache
* intellectual/mental retardation
* nausea, vomiting
* patient already included in the protocol
* pain requiring immediate medical attention. analgesic (VAS >5 and described as intolerable).

Ages: 9 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: For all patients included, a data collection form must be completed, mentioning age, sex, medical and surgical history, and the type of procedure planned.
  * If initial VAS >5 and intolerable: patients will immediately use painkillers and will be excluded from the study.
  * If initial VAS<=5 or > 5 but tolerable: Only VR glasses are used as an analgesic.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
frequency of success | 30 minutes
  frequency of success (%) (use of emergency analgesics)

SECONDARY OUTCOMES:
reduction of pain | 30 minutes
  reduction in pain assessed by the visual analog scale (mm)

OTHER OUTCOMES:
occurrence of adverse events and patient satisfaction | 3 hours
  occurrence of adverse events, tolerance to glasses, patient satisfaction (Likert Satisfaction Scale) and max VAS during the procedure.